CLINICAL TRIAL: NCT04960813
Title: Neurally Targeted Interventions to Reduce Early Childhood Anxiety
Brief Title: Kidpower Camp - Structured Games or Playgroup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Michigan State University (Other); University of Michigan (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Kate D. Fitzgerald, MD, Ruane Professor of Child and Adolescent Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU8442; 1R33MH121641-01A1 (NIH); NYSPI 8263 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders
Keywords: Effortful Control; Preschool; Error-related negativity
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Children will be randomized 1:1 to structured games or a playgroup. The structured games and playgroup will run in parallel.
Who Masked: Outcomes Assessor
Masking Description: The rater will be blinded to which intervention, structured games or playgroup, child participants receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kidpower - Structured Games (Experimental): Structured Games Camp.
  Interventions: Behavioral: Structured games
- Kidpower - Playgroup (Active Comparator): Playgroup camp
  Interventions: Behavioral: Playgroup

INTERVENTIONS:
Behavioral: Structured games — Camp Kidpower - Structured Games is an interactive, child-friendly "camp" and is comprised of short, game-like exercises taught by "camp counselors" to groups of approximately 4-6 children. In total, 15 different exercises will be taught. Children will attend 5 three-hour playgroup sessions over a 4-week period (twice the first week, and then only once per week for the subsequent 3-week period) to match the Playgroup intervention.
  Parents will be asked to attend an approximately one-hour group meeting, during which information is presented regarding child anxiety, effortful control and the rationale for this treatment. Parents are asked to continue to utilize the intervention at home every day if possible with the child and will receive texts or emails to track the games that are played at home.
  Arms: Kidpower - Structured Games
Behavioral: Playgroup — Camp Kidpower - Playgroup includes structured play activities. This will include art activities, dramatic play props, and a "story time". Children will attend 5 three-hour playgroup sessions over a 4-week period (twice the first week, and then only once per week for the subsequent 3-week period) to match the Kidpower intervention.
  During the first week parents will attend an approximately one-hour group meeting, during which information is presented regarding the positive benefits of child-led play and "special time" with caregivers.
  Parents well be asked to complete homework with their children during the week between sessions, and are shown how to track time spent in this activity. Parents will receive a daily text (or email) to to measure frequency of homework practice between sessions.
  Arms: Kidpower - Playgroup

SUMMARY:
Clinically significant anxiety affects 20% of preschoolers and can become chronic, leading to depression, substance abuse, school-drop out and even suicide. To reduce anxiety and prevent its sequelae, clinically affected children must be effectively treated early. Available interventions for clinically anxious preschoolers are effective for some, but not all children, with as many as 50% of 4-7 year olds continuing to meet criteria for an anxiety disorder after treatment.

This trial aims to help learn how Camp Kidpower, trainings using either structured games or a playgroup, may lower anxiety in preschool age children. Playing these games and learning that kids can do it, can teach kids how to keep going when they are feeling anxious. To find out if Kidpower works by helping kids stay in charge of their behaviors and emotions, the study will look at parts of the brain as well as behaviors related to effortful control and fear, before and after training.

The study hypothesizes that Kidpower will produce greater increases in Error-related negativity (ERN), Interchannel Phase Synchrony (ICPS) and effortful control (EC) behaviors than in the Playgroup control.

ELIGIBILITY:
Inclusion Criteria:

1. Children between ages 4 -5.99 years at time of consent
2. Children that have a primary clinical diagnosis of separation anxiety disorder, social anxiety disorder, generalized anxiety disorder, panic disorder, and/or obsessive-compulsive disorder
3. Written informed consent by a parent/legal guardian and verbal assent from participant
4. Fluent in English

Exclusion Criteria:

1. History of head injury
2. History of serious medical or neurological illness
3. History of post-traumatic stress disorder (PTSD)
4. History of major depressive disorder (MDD)
5. Current psychotherapy or behavioral interventions
6. History of Neurodevelopmental delay, autism spectrum disorder (ASD), or intellectual disability
7. Currently taking medications that affect central nervous system functioning
8. Primary clinical diagnosis is selective mutism or specific phobia
9. Recent history of physically aggressive behaviors that have caused harm to other children
10. Sibling of a child who has participated or is currently participating in this protocol

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate D Fitzgerald, M.D., Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Columbia University, New York, New York
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The numbers in the Participant Flow represent individual participants.
Pre-assignment Details: Participants complete a clinical assessment that determines eligibility. Of the 158 participants, 26 were ineligible from assessment, and 22 withdrew or were not responsive, leaving 110 randomized to treatment.
Groups:
- Kidpower - Structured Games: Structured Games Camp.
  Structured games: Camp Kidpower - Structured Games is an interactive, child-friendly "camp" and is comprised of short, game-like exercises taught by "camp counselors" to groups of approximately 4-6 children. In total, 15 different exercises will be taught. Children will attend 5 three-hour playgroup sessions over a 4-week period (twice the first week, and then only once per week for the subsequent 3-week period) to match the Playgroup intervention.
  Parents will be asked to attend an approximately one-hour group meeting, during which information is presented regarding child anxiety, effortful control and the rationale for this treatment. Parents are asked to continue to utilize the intervention at home every day if possible with the child and will receive texts or emails to track the games that are played at home.
- Kidpower - Playgroup: Playgroup camp
  Playgroup: Camp Kidpower - Playgroup includes structured play activities. This will include art activities, dramatic play props, and a "story time". Children will attend 5 three-hour playgroup sessions over a 4-week period (twice the first week, and then only once per week for the subsequent 3-week period) to match the Kidpower intervention.
  During the first week parents will attend an approximately one-hour group meeting, during which information is presented regarding the positive benefits of child-led play and "special time" with caregivers.
  Parents well be asked to complete homework with their children during the week between sessions, and are shown how to track time spent in this activity. Parents will receive a daily text (or email) to to measure frequency of homework practice between sessions.
Period: Overall Study
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
Started | 57 | 53
Completed | 49 | 44
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We could not retrieve the ages of 4 participants due to destroyed paperwork for de-identification purposes.
  years
    number analyzed (Participants) | 56 | 50 | 106
    (all) | 4.45 (0.50) | 4.46 (0.54) | 4.45 (0.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 21 | 61
  Male | 17 | 32 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 46 | 39 | 85
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 5 | 7
  White | 33 | 30 | 63
  More than one race | 15 | 9 | 24
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 53 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change in Error Related Negativity (ERN)
Description: The error-related negativity is a neurophysiological signal, measured via electroencephalogram (EEG), considered to reflect a dorsal anterior cingulate cortex (ACC) response to errors. For this study the ERN will be measured at electrode site FCz as the downward (negative voltage) deflection of the EEG signal that occurs 50-100 msec after error commission on the Zoo Task. Scores are measured continuously (no established minimum or maximum) . Higher scores reflect greater neural capacity for effortful control.
Time Frame: Pre-treatment (baseline) and post-treatment assessments (approximately 4-6 weeks)
Population: 18 participants from structured games and 12 participants from playgroup did not complete pre or post camp EEG or did not yield usable EEG data.
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
Number analyzed (Participants) | 31 | 32
millivolts | -0.169 (8.129) | -1.192 (10.194)

2. Primary Outcome: Change in National Institutes of Health (NIH) Toolbox Effortful Control (EC) Composite Scale
Description: The NIH Toolbox EC Composite Scale will be comprised of children's standardized scores reflecting accuracy and reaction time on two computerized tasks: the Flanker inhibitory control and attention task and the Dimensional Change Card Sort (DCCS) test of set-shifting function. An NIH Toolbox EC Composite score will be based on factor loadings for each task derived from a factor analysis of scores across both Toolbox tasks. Scores are measured continuously (no established minimum or maximum) . Higher scores reflect greater behavioral capacity for effortful control.
Time Frame: Pre-treatment (baseline) and post-treatment assessments (approximately 4-6 weeks)
Population: 5 participants from structured games and 1 participant from playgroup did not complete the NIH toolbox or did not yield usable data at pre and/or post camp visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
Number analyzed (Participants) | 44 | 43
score on a scale | .3265 (.628) | .406 (.5655)

3. Primary Outcome: Change in Clinical Global Impressions -Severity and Improvement Scales
Description: The Clinical Global Impressions (CGI) is an observer rated scale used to assess anxiety severity (CGI-S) and pre- to post-treatment improvement in anxiety (CGI-I). Ratings for both use a 7-point scale, from 1 "normal" to 7 "among the most severely ill" for CGI-S and 1 ("very much improved") to 7 ("very much worse") for CGI-I.
Time Frame: Pre-treatment (baseline) and post-treatment assessments (approximately 4-6 weeks)
Population: Of the 93 completers, 2 participants did not complete the post-camp CGI-S/I. An additional 4 CGI-S/I were unavailable for analysis, leaving 87 CGI-S/I for the final analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
Number analyzed (Participants) | 45 | 42
score on a scale
  CGI-S | 1.16 (0.93) | 1.14 (0.98)
  CGI-I | 2.44 (0.76) | 2.67 (0.87)

4. Secondary Outcome: Change in Anxiety Disorders Interview Schedule - Parent Version (ADIS-P)
Description: ADIS-P is a semi-structured clinical interview administered to parents about their child to assess Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnoses where anxiety is a component. Severity of symptoms is rated by interviewers on a scale from none (=0) to very severe (=8), with clinician severity rating (CSR) ≥ 4 indicating presence of diagnosis. Changes in CSR of the primary (i.e., most severe at baseline) anxiety diagnosis from pre to post intervention will be assessed.
Time Frame: Pre-treatment (baseline) and post-treatment assessments (approximately 4-6 weeks)
Population: Of the 93 completers, 2 participants did not complete the post-camp ADIS. An additional 4 ADIS CSR were unavailable for analysis, leaving 87 ADIS CSR for the final analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
Number analyzed (Participants) | 45 | 42
score on a scale | 2.04 (1.56) | 1.94 (1.91)

5. Secondary Outcome: Change in Spence Preschool Anxiety Scale (Spence PAS)
Description: The Spence PAS is a validated instrument for the measurement of parent report of anxiety symptoms in young children. Spence PAS scores will provide a continuous rating of anxiety symptoms from 0 to 112; high scores reflect greater anxiety.
Time Frame: Pre-treatment (baseline) up to post-treatment assessments (approximately 4-6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
Number analyzed (Participants) | 49 | 44
units on a scale | -10.4 (11.4) | -6.05 (14.9)

ADVERSE EVENTS:
Time Frame: 3 months.
Arm/Group | Kidpower - Structured Games | Kidpower - Playgroup
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53
Other Adverse Events (participants affected / at risk) | 0/57 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04960813/Prot_SAP_000.pdf